CLINICAL TRIAL: NCT07377994
Title: A Prospective, Randomized, Double-blinded, Placebo-controlled Parallel Group-Clinical Trial Assessing Gut Health and Immunomodulatory Effects of Bacillus Coagulans Based Product in Healthy Adults
Brief Title: To Evaluate the Effect of Bacillus Coagulans Based Product in Gut Health and Immunomodulatory Effect in Healthy Adults
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Bioagile Therapeutics Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: BSP-25-073
Record Dates: First submitted 2026-01-05; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Healthy Subjects (HS)
Keywords: Gut health and immunomodulatory effect
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (Experimental): Probiotic
  Interventions: Dietary Supplement: Probiotic (Bacillus Coagulans)
- Arm II (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic (Bacillus Coagulans) — Experimental
  Arms: Arm I
Other: Placebo — Placebo
  Arms: Arm II

SUMMARY:
This randomized, double-blind, placebo-controlled clinical trial is designed to evaluate the effects of a Bacillus coagulans-based probiotic product on gut health, immunological parameters, and overall tolerability in healthy adult participants. The study aims to generate clinical evidence on the role of Bacillus coagulans in maintaining intestinal homeostasis and modulating immune responses under normal physiological conditions.

Gut health will be assessed through both objective and subjective measures. Intestinal inflammation will be evaluated by measuring fecal calprotectin levels, a well-established biomarker of gut mucosal inflammation. Changes in fecal calprotectin from baseline to the end of the intervention period will be compared between the probiotic and placebo groups to determine the impact of the investigational product on gut inflammatory status.

The immunomodulatory effects of the study product will be evaluated by analyzing changes in selected immune and inflammatory markers, including immunoglobulins (IgA, IgG, and IgM). These parameters will be measured at baseline and at the end of the study to assess systemic immune responses associated with supplementation and to compare outcomes between the intervention and placebo groups.

In addition to laboratory-based assessments, participant-reported outcomes related to gut health and immune status will be captured using validated questionnaires, including the Gut Health Status Questionnaire (GHSQ) and the Immune Status Questionnaire (ISQ). These tools will be used to evaluate perceived overall relief and changes in gastrointestinal and immune-related well-being over the course of the study.

Safety and tolerability of the Bacillus coagulans-based product will be evaluated throughout the study duration by monitoring adverse events and other safety parameters in both the intervention and placebo groups, ensuring suitability of the product for use in a healthy population.

Participants will be instructed to consume the assigned study product twice daily, once in the morning and once in the evening after meals, for the duration of the intervention period. Compliance with study product intake will be documented by participants in a subject diary.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged between 18 and 50 years.
2. Female participants are either not of childbearing potential, or females of childbearing potential agree to use a medically approved method of birth control and have a negative urine pregnancy test result.
3. In good general health, as determined by medical history, laboratory analysis, and physical examination performed by the study physician.
4. Willing to provide fecal samples as per the study requirements.
5. Willing to participate voluntarily and provide written informed consent.

Exclusion Criteria:

1. Women who are pregnant or lactating.
2. Subjects who are taking Antibiotic treatment.
3. Subjects suffering from Gastrointestinal disease.
4. Subjects suffering from Diabetes.
5. Subjects suffering from Chronic/iatrogenic Immunodeficiency.
6. Subjects suffering from Abnormal blood pressure.
7. Subjects who are allergic to ingredients of the study Product.
8. Subjects who are Smoker or alcoholic.
9. Subjects who have participated prior in conflicting clinical trial or have participated in the trial over the last 3months.
10. Women who are pregnant, breastfeeding, or planning to become pregnant.
11. Daily use of supplements that contain probiotics or prebiotics within 30 days prior to screening or during study.
12. Subjects with medical conditions affecting immune status (e.g., rheumatoid arthritis, heart failure, hepatitis C, HIV) or taking medications that may impact the immune system, such as antibiotics, antimicrobials, or probiotic sachets.
13. Any surgical treatment within the previous three months or planned during the study.
14. Any subject, in the principal investigator's opinion, not considered suitable for enrolment.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-09-10 (Actual); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-05-10 (Estimated)

PRIMARY OUTCOMES:
Change in fecal calprotectin levels from baseline to the end of the study, | Baseline to Week 8 (or end of study)]
  Fecal calprotectin concentration (µg/g) will be measured at baseline and at the end of the study. The change from baseline will be analyzed.

SECONDARY OUTCOMES:
Changes in immunological markers (IgA, IgG, IgM) between baseline to the end of study | Baseline to week 8 (end of the study)
  Immunological markers (IgA, IgG, IgM) will be measured at baseline and at the end of the study. The change from baseline will be analyzed
Change in Gut Health Status Questionnaire (GHSQ) Total score from baseline to End of the Study | Baseline to week 8 (End of the Study)
  The Gut Health Status Questionnaire (GHSQ) Total score will be assessed at the baseline and at the end of the study. The change from baseline will be analyzed
Change in Immune Status Questionnaire (ISQ) Total Score from Baseline to End of the Study | Baseline to week 8 (End of the Study)
  The Immune Status Questionnaire (ISQ)total score will be assessed at the Baseline and at the end of the study. The change from Baseline will be analyzed

CONTACTS AND LOCATIONS:
Overall Officials: Parag Saudagar, Study Director — S K Biobiz Private Limited
Locations (1):
- Advanced Gastro Care, Bangalore, Karnataka, India

IPD SHARING:
Plan to Share IPD: No